CLINICAL TRIAL: NCT04230837
Title: Marginal Bone Levels Around Implants With Definitive Abutments Of One and Three Millimeters: A One Year Of Follow Up Randomized Clinical Trial
Brief Title: Marginal Bone Level Around Implants With Definitive Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jose Nart Molina, Chairman and Program Director, Department of Periodontology at UIC Barcelona, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2015-05
Record Dates: First submitted 2019-11-18; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Implant Site Reaction
Keywords: definitive implant abutment; interproximal bone loss; soft tissue

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective study
Who Masked: Participant
Masking Description: The surgeon was unaware of the abutment height until after the insertion of the implant. Patients were unknown the abutment group. The examiner, independent to the study, carried out the radiographic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Abutments of 1 mm (Experimental): Definitive abutments of 1 mm height were located.
  Interventions: Device: Inmediate abutment height
- B: Abutments of 3 mm (Experimental): Definitive abutments of 3 mm height were located.
  Interventions: Device: Inmediate abutment height

INTERVENTIONS:
Device: Inmediate abutment height — The placement of the implant was done following the manufacturing protocol and using a surgical guide according to the radiological guide previously used. At this time, the Permanent® abutment of 1 or 3 mm was chosen randomly and was placed at 35 Ncm.

SUMMARY:
The aim of the present study was to evaluate the peri-implant crestal bone level around implants placed 1.5 mm subcrestally, with a 1 mm or 3 mm definitive abutment height at the time of implant placement after 1 year. Patients were selected from the Department of Periodontology at Universitat Internacional de Catalunya. X-rays were taken at the time of implant placement, 8-12 weeks after placement, after screwing the provisional rehabilitation and at 12 months. An examiner indicated the crestal marginal bone level, the marginal bone level of the implant, and the marginal bone level of the abutment . The examiner, independent to the study, carried out the radiographic analysis using the Image J software on periapical radiographs.

DETAILED DESCRIPTION:
The aim of the present study was to evaluate the peri-implant crestal bone level around implants placed 1.5 mm subcrestally with PS and a 1 mm or 3 mm definitive AH at the time of implant placement after 1 year.

1. Study design

   This randomized controlled prospective study was carried out after its acceptance by the Clinical Research Ethics Committee with code number PER-ECL-2015-05, at the Faculty of Dentistry of the Universitat Internacional de Catalunya (UIC-Barcelona).
2. Study population and selection criteria

   Patients were selected from the Department of Periodontology at Universitat Internacional de Catalunya. Once signed the informed consent, patients were screened following inclusion criteria.
3. Randomization

   The randomization between the groups (Group A/Group B) was performed using OxMaR system (Oxford Minimization and Randomization) to determine the use of a 1 mm (Group A) or 3 mm (Group B) height abutments. The surgeon was unaware of the abutment height until after the insertion of the implant.
4. Surgical and prosthetic treatment protocol Dental implants were placed by second and third year students of the Postgraduate Program in Periodontology at UIC-Barcelona, supervised by two experienced professors (MM, MA). Vega® implant, Klockner, several lengths (8, 10, 12 mm) and diameters (3.5, 4.0, 4.5 mm) were used depending on bone availability. The rehabilitation was carried out by students of the Postgraduate program of Esthetic and Prosthetic Dentistry at UIC-Barcelona, using the permanent prosthetic abutments with two different heights (1 or 3 mm) placed the day of surgery. The screwed-retained rehabilitations to the Permanent® abutment were single crowns or partial restorations (maximum of 3 crowns), both performed with CAD-CAM technology. Temporary restorations were placed between 2 to 4 months after surgery, for 4 weeks, before the placement of the definitive ones.

   Treatment sequence:
   * Preparation and implant surgery: a radiologic guide on a CBCT scan, and a standardized periapical radiograph were made for every patient. Pre-surgical instructions and medication such as antibiotic prophylaxis was made with 500 mg Amoxicillin every 8 h starting 1 hour prior to surgery, and 500mg/8h for 7 days. In allergic patients, Clindamycin 300 mg every 8 h, starting 1 day previously was used, and 300mg/8h/7days. The KM thickness was assessed before raising the mucoperiosteal flap. The placement of the implant was done following the manufacturing protocol and using a surgical guide according to the radiological guide previously used. IAll implants were placed 1.5 mm subcrestally from the most apical area of the crest, using a periodontal probe. At this time, the Permanent® abutment of 1 or 3 mm was chosen randomly and was placed at 35 Ncm. Postoperative anti-inflammatory medication (ibuprofen 600 mg, 1 tablet / 8 h / if pain) and 0.12% chlorhexidine rinse (2 times / day / 7 days) were advised. A standardized periapical radiograph was performed immediately after the implant placement. The amount of Keratinized gingiva (KG) was recorded and also the stability values of the implant by using the Penguin® device (RFA values) to the implant and on the Permanent abutment.
   * Prosthetic treatment: After 10 weeks up to 4 months, impressions were taken with fluid and heavy silicone (Zhermack® elite HD +) to make the provisional prosthesis, as long as the RFA values were greater than 65 ISQ. At the time of the temporary resin prosthesis placement, all the following clinical parameters (PD, mPI, mSBI, KG, BG, S, POI) were recorded and a periapical radiograph also taken. The definitive prosthesis was performed 4 weeks after the placement of the provisional. Records of clinical measures (BG, MT, mPII, mSBI, PD, KM) and periapical X-ray (periapical). clinical follow-up (MT, mPII, mSBI, PD), radiographic (periapical and orthopantomography) and RFA were evaluated 12 months later.
5. Radiographic evaluation X-rays were taken at the time of implant placement, 8-12 weeks after placement, after screwing the provisional rehabilitation and at 12 months. Radiographs were standardized by using an individualized radiographic stent for each patient, thus ensuring a parallel technique. (Figure 1 and 2) MBL measurements were performed by one examiner who recorded on each radiograph mesially and distally, the most coronal part of the bone crest (C), the position of the implant shoulder (H), and the level of the first peri-implant bone contact with the implant (Fi ) or abutment (Fa). Then, the examiner measured the distance in millimeters of H-C, which defined the crestal marginal bone level (MBLc), while the shoulder distance of Fi was the marginal bone level of the implant (MBLi). When the first contact was located in the abutment, the distance H and Fa was recorded as the marginal bone level of the abutment (MBLa). The distance MBLc was considered positive if the mark C was coronal to H, negative if C was apical, and zero if Fi and H coincided (Figure 3). The changes in MBLc (CMBLc) were registered at 12 months with respect to the baseline. Changes in MBLc, MBLi or MBLa (CMBLc, CMBLi, CMBLa) were measured in the same time period at 12 months.
6. Calibration The examiner, independent to the study, carried out the radiographic analysis using the Image J software (Java image processing program by Wayne Rasband; National Institutes of Health (NIH), USA) on periapical radiographs, with a x7 magnification. Previously, the examiner was calibrated 3 times separately, with an interval of 72 hours, making measurements at 10 radiographs to determine the intraoperator reproducibility. The aim was to obtain an intraclass coefficient of 0.99 (P <.05) as the intraoperator reliability coefficient.
7. Stability evaluation The resonance frequency analysis, RFA was recorded with the Penguin® system (Integration Diagnostics Sweden) at the time of implant placement, 10-12weeks and 1year.
8. Sample size Accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a bilateral contrast, 28 subjects were required in each group to detect a difference equal to or greater than 0.5mm. It was assumed that the standard deviation (SD) was 0.59 and a possible drop-out of 20% was estimated.
9. Statistical analysis Analysis was performed at implant level. In order to describe the qualitative variables, absolute frequencies and percentages were used. The description of quantitative variables was performed using the mean and SD. Normal distribution of each parameter was assessed by the Shapiro-Wilk test, and as data did not follow a normal distribution a Wilcoxon test was used to compare interproximal MBLs between baseline and 12 months follow-up, and Mann-Whitney U-test was used to compare interproximal MBL changes between treatment groups. The level of statistical significance was set at p < 0.05. The statistical package SPSS 22.0 (IBM, SPSS, SPSS Inc., Chicago, IL, USA) was used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old;
* Controlled ASA1 or ASA2 patient;
* Healthy periodontium or with controlled periodontal disease;
* Need for rehabilitation with implants in partially posterior edentulous sextants;
* Full Mouth Plaque Score (FMPS) less than 20% at the time of surgery;
* Collaborating patients.

  * According to the implant location:
* Healed posterior sites, with a minimum of 2 months post-extraction;
* Ridge width of 7 mm or more and of 10 mm of height to the mandibular nerve and 8 mm to the maxillary sinus;
* Minimum keratinized mucosa (KM) width of 4 mm;
* Antagonist dentition having a fixed restoration or natural teeth, (5) restorative space greater than 5 mm.

Exclusion Criteria:

* Patients with endocrine, immunological or metabolic alterations;
* Pregnancy, allergy to any metallic component of the implant;
* Drug consumption or alcoholism;
* Tobacco ≥10 cig/d and
* Severe bruxism and TMJ pathology.

  * According to the implant location:
* Require regeneration techniques;
* Width of KM less than 2 mm at any implant site;
* Infections in the treatment area;
* Absence of implant primary stability and
* Being unable to perform prosthetically guided screw-retained restorations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Bone Loss, at 8-12 weeks and 1 year. | baseline, 8-12 weeks and 1 year
  X-rays were taken at the time of implant placement, 8-12 weeks after placement, after screwing the provisional rehabilitation and at 12 months.
Mucosal thickness (MT) | baseline
  Mucosal thickness (MT) before placement of the implant using a PCP-UNC15 periodontal probe. This measure will be compared with the abutment high and bone loss at 1 year.

SECONDARY OUTCOMES:
Change from Baseline the resonance frequency analysis at 8-12 weeks and 1 year. | baseline, 8-12 weeks and 1 year
  RFA was recorded with the Penguin® system at the time of implant placement, 8-12weeks and 1 year later.
Plaque index at 1 year | 1 year
  Plaque index (mPII, modified plate index, Mombelli et al., 1987)
Bleeding on probing at 1 year | 1 year
  Presence of bleeding on probing (mSBI, Modified bleeding index, Mombelli et al., 1987)
Probing depth at 1 year | 1 year
  Probing depth (PD) (6 locations MV / V / DV / MP / P / DP): with a periodontal probe PCP-UNC15;

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco J, Pico A, Caneiro L, Novoa L, Batalla P, Martin-Lancharro P. Effect of abutment height on interproximal implant bone level in the early healing: A randomized clinical trial. Clin Oral Implants Res. 2018 Jan;29(1):108-117. doi: 10.1111/clr.13108. Epub 2017 Dec 8. PMID 29222809
- [Background] Borges T, Leitao B, Pereira M, Carvalho A, Galindo-Moreno P. Influence of the abutment height and connection timing in early peri-implant marginal bone changes: A prospective randomized clinical trial. Clin Oral Implants Res. 2018 Sep;29(9):907-914. doi: 10.1111/clr.13343. PMID 30259582
- [Background] Chen Z, Lin CY, Li J, Wang HL, Yu H. Influence of abutment height on peri-implant marginal bone loss: A systematic review and meta-analysis. J Prosthet Dent. 2019 Jul;122(1):14-21.e2. doi: 10.1016/j.prosdent.2018.10.003. Epub 2019 Feb 16. PMID 30782461
- [Background] Galindo-Moreno P, Leon-Cano A, Ortega-Oller I, Monje A, Suarez F, OValle F, Spinato S, Catena A. Prosthetic Abutment Height is a Key Factor in Peri-implant Marginal Bone Loss. J Dent Res. 2014 Jul;93(7 Suppl):80S-85S. doi: 10.1177/0022034513519800. Epub 2014 Mar 12. PMID 24621670
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. Reaction of crestal bone around implants depending on mucosal tissue thickness. A 1-year prospective clinical study. Stomatologija. 2009;11(3):83-91. PMID 19996674
- [Background] Linkevicius T, Puisys A, Steigmann M, Vindasiute E, Linkeviciene L. Influence of Vertical Soft Tissue Thickness on Crestal Bone Changes Around Implants with Platform Switching: A Comparative Clinical Study. Clin Implant Dent Relat Res. 2015 Dec;17(6):1228-36. doi: 10.1111/cid.12222. Epub 2014 Mar 28. PMID 24673875
- [Background] Molina A, Sanz-Sanchez I, Martin C, Blanco J, Sanz M. The effect of one-time abutment placement on interproximal bone levels and peri-implant soft tissues: a prospective randomized clinical trial. Clin Oral Implants Res. 2017 Apr;28(4):443-452. doi: 10.1111/clr.12818. Epub 2016 Mar 25. PMID 27016157
- [Background] Novoa L, Batalla P, Caneiro L, Pico A, Linares A, Blanco J. Influence of Abutment Height on Maintenance of Peri-implant Crestal Bone at Bone-Level Implants: A 3-Year Follow-up Study. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):721-727. doi: 10.11607/prd.2762. PMID 28817138
- [Background] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250
- [Background] Spinato S, Stacchi C, Lombardi T, Bernardello F, Messina M, Zaffe D. Biological width establishment around dental implants is influenced by abutment height irrespective of vertical mucosal thickness: A cluster randomized controlled trial. Clin Oral Implants Res. 2019 Jul;30(7):649-659. doi: 10.1111/clr.13450. Epub 2019 May 12. PMID 31033035
- [Background] Vervaeke S, Dierens M, Besseler J, De Bruyn H. The influence of initial soft tissue thickness on peri-implant bone remodeling. Clin Implant Dent Relat Res. 2014 Apr;16(2):238-47. doi: 10.1111/j.1708-8208.2012.00474.x. Epub 2012 Jul 3. PMID 22758656
- [Background] Canullo L, Camacho-Alonso F, Tallarico M, Meloni SM, Xhanari E, Penarrocha-Oltra D. Mucosa Thickness and Peri-implant Crestal Bone Stability: A Clinical and Histologic Prospective Cohort Trial. Int J Oral Maxillofac Implants. 2017 May/June;32(5):675-681. doi: 10.11607/jomi.5349. Epub 2017 Mar 15. PMID 28296981